CLINICAL TRIAL: NCT06557070
Title: The Effect of Emotional Freedom Technique on Premenstrual Syndrome, Menstrual Symptom and Life Quality of Nursing Students: A Randomized Controlled Study
Brief Title: The Effect of Emotional Freedom Technique on Premenstrual Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hande Yagcan, Associate Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DokuzEU_THEFT
Record Dates: First submitted 2024-07-19; First posted 2024-08-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Premenstrual Syndrome; Emotional Freedom Technique; Nursing Caries
Keywords: Premenstrual Syndrome; menstrual symptom; life quality; emotional freedom technique; Nursing Care
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled experimental study
Who Masked: Participant
Masking Description: To ensure blinding in the study, randomization will be carried out by someone other than the researchers. A total of 8 sessions of Emotional Freedom Technique (EFT) will be applied to the experimental group, once a week. No application other than the scales will planned for the control group. Only, the control group will be taught the EFT technique at the end of the experiment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emotional Freedom Technique (EFT) experimental group (Experimental): A total of 8 sessions of Emotional Freedom Technique (EFT) will be applied to the experimental group, once a week. First, the experimental group was informed about premenstrual syndrome and EFT face to face and EFT application was taught. EFT application was performed every week for 2 cycles. During the application, plans were made to be face-to-face, online, in a group or individually. The posttest was repeated after the application was completed.
  Interventions: Other: The Emotional Freedom Technique
- The control group. (No Intervention): The control group was first given a pre-test, then given information about premenstrual syndrome face to face, no intervention was made, they were asked not to use painkillers, a post-test was performed at the end of 2 cycles, and EFT was taught to the students who wanted it.

INTERVENTIONS:
Other: The Emotional Freedom Technique — Emotional freedom technique (EFT) is a method to help manage emotions and troubling thoughts and lower stress and anxiety. EFT is applying by tapping. To do EFT, you tap your fingertips on certain points on your hand, head, and torso which are used in acupuncture.
  Arms: Emotional Freedom Technique (EFT) experimental group

SUMMARY:
Introduction: Premenstrual Syndrome (PMS) is a condition that occurs in the luteal phase of the menstrual cycle and affects women's lives physically, psychologically and behaviorally, starting approximately five days before menstruation and decreasing spontaneously a few days later.

Purpose: This research is planned to examine the effect of the Emotional Freedom Technique on the experience of premenstrual syndrome and menstrual symptoms and the quality of life of nursing students with premenstrual syndrome.

Method: The research will be conducted with first, second, third and fourth year female students studying at Dokuz Eylül University Faculty of Nursing. Diagnostic information form, premenstrual syndrome scale, menstruation symptom scale, SF-12 quality of life scale and subjective danger units will be collected via Google form. SUD Scale will be applied. The research is designed with experimental and control groups, and it is found that a total of 70 female students are needed, 35 in the experimental group and 35 in the control group. PMSS analysis will be performed and students who score over 132 points and meet the inclusion criteria will be numbered in the order of filling out the survey, and randomization will be done using the "Random Sequence Generator" through www.random.org, which provides computer-assisted randomization, and experimental and control groups will be created. Simple randomization will be applied to keep the control and experimental groups equal. To ensure blinding in the study, randomization will be carried out by someone other than the researchers. A total of 8 sessions of Emotional Freedom Technique (EFT) will be applied to the experimental group, once a week. No application other than the scales will planned for the control group.

DETAILED DESCRIPTION:
Premenstrual Syndrome (PMS) is a condition that occurs during the luteal phase of the menstrual cycle and begins approximately five days before menstruation, subsiding spontaneously a few days later. It affects women's lives physically, psychologically, and behaviourally. PMS is a common health issue among menstruating women, with a has a global prevalence of 47.8%, while its prevalence in Turkey is 52.2%. Although the exact aetiology of PMS is unknown, it is thought to be influenced by factors such as excess or deficiency of oestrogen, aldosterone and renin-angiotensin imbalance, progesterone deficiency, and thyroid dysfunction.

The Emotional Freedom Technique (EFT) is used to improve conditions such as anger, sadness, anxiety, and depression, where the individual's physical or psychological awareness is focused on a specific issue. EFT is based on the existence of an energy system (meridian system) that surrounds the physical body like a network. It involves tapping, pressing, and stimulating selected acupuncture points, particularly on the head and upper body, using the fingertips along these meridians. While applying pressure with the fingertips, a specific phrase related to the problem is recited. Each point is tapped at least seven times. Completing the specific phrase and taps is called an 'EFT round'.

A review of the literature reveals that PMS and its symptoms negatively impact women's lives in physical, psychological, and behavioural terms. This negative impact is also thought to adversely affect the individual's comfort and reduce their quality of life. As a coping method, EFT is effective in managing symptoms due to its low cost, reliability, absence of side effects, and ease of self administration. According to Clond (2016), more studies are needed to determine the effectiveness and level of evidence of EFT. This need can be met by increasing the number of randomised controlled trials and meta-analyses. This need can be met by increasing the number of randomised controlled trials and meta-analyses. We anticipate that our study, which was initiated for this purpose, will contribute to both the literature and practice. Furthermore, a review of the literature reveals that education, acupressure, and yoga methods are commonly used in studies on coping with PMS. One RCT study using the EFT method was found, but there was a lack of clarity on issues such as on which day of the menstrual cycle EFT was started, who performed the application, and whether the students performed the application or not. Differences were also found between the scales used in that study and our study. In this study, our aim is to improve the quality of life of nursing students experiencing PMS by reducing their premenstrual syndrome and menstrual symptoms through the application of EFT.

Inclusion Criteria;

* Scoring 132 or above on the Premenstrual Syndrome Scale (achieving 50% of the scale's total points),
* Aged 18 years or older,
* With a menstrual cycle length within normal limits (every 21-35 days) for the past three months,
* Voluntarily participating in the study,
* Possessing a smartphone and internet access, female students were included.

Exclusion Criteria:

* Receiving psychiatric treatment,
* Having started antidepressants in the last three months,
* Using oral contraceptives were excluded from the study. The G.Power 3.1 programme was used to determine the numbers of the experimental and control groups for the study. The calculation was made by referring to the study by Bakır, Irmak Vural and Körpe (2021) and 35 experimental groups and 35 control groups, totalling 70 students, were calculated at 80% power and 95% confidence interval.

To prevent potential data loss, 80 female students who met the inclusion criteria were grouped into 40 experimental and 40 control groups.

In an experimental study, keeping losses below 10% or 15% is considered important in reducing bias, and it is emphasised that increasing the sample size is useful in controlling bias associated with losses.

The groups included in the study were divided into two groups: the experimental group and the control group. A simple random method was used to select participants for the study. The pre-test measurements of the participants to be included in the study were collected by the researchers, and an independent statistician assigned IDs and sequence numbers to the relevant individuals. The experimental and control groups were determined blindly by an independent statistician using a lottery. The randomisation results obtained using Randomizer.org . The students included in the study did not know which group they were in. Furthermore, the analysis of the study was conducted by an independent statistician. The study is registered on ClinicalTrials.gov (Id No: NCT06557070). The study was conducted according to the Updated Guidelines for Reporting Randomised Parallel Group Studies (Consolidated Standards of Reporting Trials-CONSORT).

ELIGIBILITY:
Inclusion Criteria:

* Scoring over 132 on the premenstrual syndrome scale
* Over 18 years old
* Having had a regular menstrual cycle for the last three months (21-35)
* Owner of a smartphone and internet
* Agreeing to participate in the research

Exclusion Criteria:

* Psychiatric treatment and antidepressant medication in the last three months who have started,
* Who are pregnant,
* Who have given birth,
* Who use oral contraceptives,
* Who have difficulty accessing the internet
* Who did not participate in the post-test will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Premenstrual syndrome is a disorder that affects women and especially adolescent girls, reducing their quality of life and negatively affecting their educational achievement and work life. Reducing these symptoms is a positive attempt to empower women.
Enrollment: 70 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | Before the EFT application
  The Personal Information Form is a form consisting of 22 questions regarding socio-demographic characteristics, lifestyle and menstrual history, created by the researcher using the relevant literature in order to obtain the data of the female students to be included in the research and to perform randomization effectively.

SECONDARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | Before and 3 months after the EFT application trial
  It is a scale that aims to describe premenstrual symptoms and measure the severity of symptoms. Answers to the items on the scale are marked taking into account the situation of "being within the week before menstruation" as stated in the instructions. Scale, depressive affect , anxiety , fatigue , irritability , depressive thoughts , pain , appetite changes , It consists of nine subscales: sleep changes and bloating . The scale score is determined by the score obtained from the sub-dimensions. This score is called the "PMSÖ total score" and the lowest score that can be obtained is 44 and the highest score is 220. Increasing the scale score means increasing symptoms.

OTHER OUTCOMES:
Menstruation Symptom Scale (MSS) | Before and 3 months after the EFT application trial
  It was developed to evaluate menstrual pain and symptoms. Participants are asked to give a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. 1-13. Items belong to the "Negative effects/somatic complaints" subscale, items 14-19. The items refer to the "Menstrual pain symptoms" subscale and items 20-22. The items belong to the "Coping methods" sub-dimension. It is a five-point Likert type scale consisting of 22 items. The score obtained from the sub-dimensions is calculated by taking the total score average of the items in the sub-dimensions. An increase in the mean score for sub-dimensions indicates that the severity of menstrual symptoms related to that sub-dimension has increased.
Subjective Units of Distress Scale (SUDS) | Before and 3 months after the EFT application trial
  During the subjective evaluation, the individual considers the discomfort he/she feels in response to the stimulus that causes his/her anxiety as "0" as "no discomfort" and "10" as "unbearable discomfort" and scores his/her discomfort on a scale between 0-10. A high score means that the level of anxiety or stress felt by the individual is high.

CONTACTS AND LOCATIONS:
Overall Officials: Hande Yagcan, Assoc Prof, Study Director — Dokuz Eylul University Faculty of Nursing
Locations (1):
- Dokuz Eylul University Faculty of Nursing, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No